CLINICAL TRIAL: NCT04998513
Title: Medical Versus Surgical Treatment for Peritonsillar Abscesses: a Pilot Study for a Randomized, Multi-institutional Pragmatic Superiority Trial
Brief Title: Medical Versus Surgical Treatment for Peritonsillar Abscesses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This project was never submitted or reviewed by the NSH REB; reason unknown
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23821
Record Dates: First submitted 2020-06-23; First posted 2021-08-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Peritonsillar Abscess; Surgical Incision
MeSH Terms: conditions — Peritonsillar Abscess; Surgical Wound

STUDY DESIGN:
Intervention Model Description: The proposed trial is designed as a randomised, controlled, analyst blinded, multi-institutional, pragmatic superiority trial with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: Analysts will be masked as to the study arm participants are randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Management Alone Arm (Active Comparator): Antibiotics, steroids, fluids
  Interventions: Drug: Medical Management Alone Arm
- Surgical Arm (Active Comparator): Incision and drainage
  Interventions: Procedure: Surgical Arm

INTERVENTIONS:
Drug: Medical Management Alone Arm — The medical intervention consists of intravenous dexamethasone (10 mg if bodyweight < 70 kilograms, 20 mg if bodyweight > 70 kilograms), intravenous cefazolin 2 grams, intravenous metronidazole 500 mg, oral probenecid 2 grams, and 1 liter of intravenous crystalloid fluid given over 1 hour.
  If, during the initial post-enrolment day 1 follow-up, patients report a failure of signs and symptoms to improve since their medical therapy, a second round of intravenous crystalloid fluid, cefazolin, probenecid, metronidazole and dexamethasone will be given at the same dose as the initial medical therapy. Failure to improve patient signs and symptoms over a two-hour observation window will prompt surgical intervention to be performed in the same fashion as the surgical intervention group.
  Arms: Medical Management Alone Arm
Procedure: Surgical Arm — Surgical intervention consists of attempted incision and drainage of the abscess. Specific procedure steps and details are at the discretion of the treating surgeon. In general, incision and drainage consists of topical and submucosal local anesthetic followed by a mucosal incision along the palatoglossal arch and soft palate junction, and blunt dissection of the abscess cavity to evacuate pus. Some surgeons may first perform a needle aspiration. For purposes of the trial, positive aspiration of pus on needle aspiration must be followed by attempted incision and drainage. Failed needle aspiration or surgical drainage will be considered as a failed attempt at surgical intervention.
  Patients randomized to receive surgical intervention will also receive medications as per the medical management arm.
  Arms: Surgical Arm

SUMMARY:
Peritonsillar abscesses are major infections around the tonsils. The abscess is a collection of pus that can cause a large amount of pain and discomfort, which can result in trouble swallowing and drinking. Peritonsillar abscesses must be treated because they can spread to other areas in the throat and neck, which can cause difficulty breathing, can even spread throughout the rest of the body.

Over the years, many different treatments have been used for peritonsillar abscesses. In the past, the entire tonsil was removed in the operating room while the patient was asleep. This surgery can cause a large amount of bleeding, and so now smaller surgeries are performed while the patient is awake. Small needles are put through the open mouth and into the abscess to drain it. As well, a small cut can be made to drain the infection. These last two treatments cause less problems than removing the whole tonsil, but there are still risks. The surgeries are uncomfortable for patients and they can cause anxiety and fear. There are also large blood vessels nearby that can be injured.

In the last few years, treatment of peritonsillar abscesses without surgery has been studied. Patients receive strong antibiotics and anti-inflammatories (known as steroids) and they may not need surgery. It is not yet known if this treatment works as well as surgery. In order to figure this out, research must look at both options compared against each other in a large study with many patients.

However, large research studies require a lot of planning, and so smaller studies are helpful to figure out if the larger study is even possible. The current study would be a small trial to plan for a larger study later on.

Patients will be randomly treated with either medications alone or with surgery. The main part of the study will look at issues with planning the future study, such as how long it takes to fill out forms, how many missing results there are at the end of the study, and how patients and doctors feel about taking part in the research study. The future large study will look at how well the treatment options reduce pain, how fast patients are able to swallow normally again, how often patients need to change treatments, and whether there are differences in quality of life with the treatment options. Because these things will be looked at in detail in the future large study, the investigators will also look at them during this small planning study, but the investigators will not be able to tell for certain which treatment is better until the large study is completed.

The results of this study are important for planning and performing the larger study, and they are important for getting future funding to do that study. Large studies are very expensive, and major funding organizations, such as the Canadian Institutes of Health Research, look for this early data when deciding who should get funding. The results of both this pilot study and the future larger study could be practice changing for how peritonsillar abscesses are treated, and will benefit both Nova Scotians and potentially the rest of world.

DETAILED DESCRIPTION:
Peritonsillar abscesses (PTA) are the most common deep neck space infection, and are amongst the most common on-call emergency consultations for otolaryngologists. The PTA is a collection of pus in the peritonsillar space resulting from untreated tonsillitis and pharyngitis. The bacteria responsible for PTA formation have fluctuated, and largely include a multitude of both anaerobic and aerobic species1,2.

Previous studies have demonstrated world-wide incidences of 10 to 40 per 100,000 people, and recent Canadian evidence has shown agreement2. Despite the tendency to be relatively benign, PTA's have potential for spread to other deep neck spaces, such as the parapharyngeal space, and can cause sepsis and airway obstruction3. The possibility of these sequelae necessitates prompt treatment of any PTA.

The diagnosis of PTA is sometimes difficult, and specific criteria are lacking. The use of radiological imaging varies geographically, and the diagnosis typically relies on clinical acumen3. However, it should be noted that the clinical spectrum between tonsillitis, peritonsillar cellulitis, and PTA can be difficult to differentiate4,5. There is no agreed upon guideline for the diagnosis and management of PTA, and current practices are unknown. Our group is currently investigating this evidence gap (study ongoing).

Management of PTA has changed over many years. Traditional approaches had previously found surgical intervention essential for treating abscesses, including combinations of needle aspiration, incision and drainage, and immediate tonsillectomy. In this regard, incision and drainage has been found to be the best option in regard to both reducing recurrence and avoiding complications such as post-tonsillectomy hemorrhage6. While surgical interventions for PTA are commonly performed procedures, they are not without risk, including the possibility of significant hemorrhage from carotid artery injury, elevated pain levels, and emotional distress7.

Given these risks, and the often-limited availability of specialist access, other authors have questioned the need for the surgical intervention of PTA. Proponents of this new approach argue that medical treatment alone results in lesser pain and faster return to normal oral intake and daily living, without an increase in treatment failure or PTA associated sequelae. Furthermore, medical treatment alone helps satisfy tenants of the Canada Health Act. A large proportion of Canada's population is rural8. While emergency surgical treatment of PTA is generally accessible through costly transportation measures such as long-distance driving, ambulance transfer, or air lift, a substantial portion of the rural population would benefit from avoidance of this transportation altogether. Regardless of its implication for policy change and accessibility, medical treatment may serve to improve patient quality of life (QOL) and patient oriented outcomes by reducing travel time and empowering non-otolaryngologist providers to competently intervene.

However, studies favoring medical treatment alone are small. Our group has recently completed a systematic review and meta-analysis of the topic9. Medical management alone was found to offer equivalent pain and oral intake outcomes with similar treatment failure rates, suggesting surgical intervention can be avoided in many patients. Studies providing evidence for medical treatment are mostly observational, with no peer-reviewed published randomized trials comparing medical and surgical treatment for PTA.

Patient reported outcomes (PRO's) such as pain and quality of life (QOL) are essential measurements for advancing care10,11. In patients with peritonsillar abscess, pain is a uniformly present symptom, and quality of life is reduced as a result of pain, inability to swallow, and multiple other factors. Removing the need for surgical intervention may reduce patient pain, anxiety, and distress without an increased risk of treatment failure. Therefore, a future clinical trial would seek to compare medical intervention alone to surgical intervention in pain reduction for uncomplicated PTA.

Pilot studies are smaller scale studies used to assess the feasibility, reliability, and validity of a proposed trial design. Results of a pilot study are used to refine or modify the design of the subsequent trial, and to assist researchers in performing a high-quality trial. Many have suggested all trials should perform an initial pilot study, both reducing potentially wasted resources and improving full trial results due to improved logistics and data efficiency12,13.

Therefore, the investigators propose a pilot study to assess the feasibility of conducting a multi-institutional, pragmatic, superiority trial investigating medical versus surgical management of adult patients with uncomplicated PTA. This pilot study will assess the process, resources, management, and scientific considerations of the proposed trial.

The proposed trial is designed as a randomised, controlled, analyst blinded, multi-institutional, pragmatic superiority trial with two parallel groups. Randomization will be via simple randomization in a balanced 1:1 ratio, with concealment and randomization by a third-party online system (Randomize.net; FDA 21 CFR Part 11 compliant).

ELIGIBILITY:
Patient inclusion criteria include:

* 1) Adult patients (> 18 years old),
* 2) Clinical diagnosis of peritonsillar abscess (with or without imaging before consultation).

Patient exclusion criteria include:

* 1) Immunocompromised state, defined as active cancer, present or recent (within 1 year) chemotherapy use, diagnosis or evidence of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS) , or diagnosis of an alternative immunodeficiency disorder
* 2) Uncontrolled diabetes mellitus, defined as random blood sugar greater than 12 millimoles per liter,
* 3) Clinical diagnosis of peritonsillar abscess extending to other deep neck spaces, defined as decreased neck range of motion, and clinical gestalt of overall illness,
* 4) Inability to handle secretions as determined by the treating clinician
* 5) Clinically severe dehydration (as determined by treating clinician's volume status assessment) or failure to thrive requiring inpatient admission,
* 6) Requirement of admission for inpatient management for any other reason,
* 7) Requirement of general anesthetic for surgical drainage,
* 8) Unable to consent to study involvement,
* 9) Patient has already received 48 hours of appropriate antibiotic coverage (below) prior to eligibility assessment.
* 10) Previous diagnosis of peritonsillar abscess (other than the current event) within the past month.

Note, the exclusion criteria of inability to handle secretions and severe dehydration are markers of severe disease that likely require surgical intervention. Patient reported dehydration or inability to handle secretions need not exclude potentially eligible patients if the treating clinician determines these factors to be clinically absent or the patient to have mild to moderate infection.

Appropriate antibiotic coverage is defined as:

1. Institutionally standard antibiotics for the treatment of peritonsillar abscess, as determined by the treating physician
2. Any of the following at appropriate dosage range:

   1. Amoxicillin-clavulanic
   2. Ceftriaxone
   3. Clindamycin
   4. Penicillin plus metronidazole
   5. Cefazolin plus metronidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 month
  The number of eligible patients screened, regardless of participation, will be recorded and compared to the number of participating patients
Retention rates | 1 month
  The number of patients completing the required follow-ups will be recorded
Compliance | 1 month
  The number of completed NPS and analgesia diaries will be recorded

SECONDARY OUTCOMES:
Burden of study involvement of both participants and investigators | 1 month
  1. Investigators will record the time at start of assessments and upon completion of assessments and related study documents
  2. Participant times will be automatically recorded by their digital collection tools, or they will record the time required on paper
  3. The time associated with recruitment documents will be examined, after-hours will be considered after 1700h
  4. Perceived burdens will be elicited during a qualitative analysis post-pilot study

OTHER OUTCOMES:
Future trial outcomes will be examined as per protocol | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Matthew H Rigby, MD MPH FRCSC, Principal Investigator — Dalhousie University, Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No